CLINICAL TRIAL: NCT00910520
Title: Botulinum Toxin Type A for the Treatment of Patients With Idiopathic Overactive Bladder With Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-520
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- onabotulinumtoxinA (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 100 U injected into the detrusor at Day 1, followed by a repeat injection of onabotulinumtoxinA 100 U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA
- placebo/onabotulinumtoxinA (Other): Placebo (normal saline) injected into the detrusor at Day 1, followed by an injection of onabotulinumtoxinA (botulinum toxin Type A) 100 U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA; Drug: normal saline

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA (botulinum toxin Type A) 100 U injected into the detrusor at Day 1, followed by a repeat injection of onabotulinumtoxinA 100 U after a minimum of 12 weeks (if applicable). Or, if placebo is administered at Day 1, onabotulinumtoxinA 100 U injected after a minimum of 12 weeks (if applicable).
  Other Names: BOTOX®; botulinum toxin Type A
Drug: normal saline — Normal saline (placebo) injected into the detrusor at Day 1.
  Arms: placebo/onabotulinumtoxinA

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of botulinum toxin type A (onabotulinumtoxinA) in treating patients with idiopathic overactive bladder with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB (frequency/urgency) with urinary incontinence for at least 6 months
* Inadequate response or limiting side effects with anticholinergics for the treatment of OAB

Exclusion Criteria:

* Overactive Bladder caused by neurological condition
* Patient has predominance of stress incontinence
* History or evidence of pelvic or urological abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (7):
- Laguna Hills, California, United States
- Ghent, Belgium
- Prague, Czechia
- Tübingen, Germany
- Warsaw, Poland
- Moscow, Russia
- London, United Kingdom

REFERENCES:
- [Derived] Castejon N, Khalaf K, Ni Q, Cuervo J, Patrick DL. Psychometric properties of the incontinence utility index among patients with idiopathic overactive bladder: data from two multicenter, double-blind, randomized, Phase 3, placebo-controlled clinical trials. Health Qual Life Outcomes. 2015 Aug 1;13:116. doi: 10.1186/s12955-015-0306-5. PMID 26231052
- [Derived] Sievert KD, Chapple C, Herschorn S, Joshi M, Zhou J, Nardo C, Nitti VW. OnabotulinumtoxinA 100U provides significant improvements in overactive bladder symptoms in patients with urinary incontinence regardless of the number of anticholinergic therapies used or reason for inadequate management of overactive bladder. Int J Clin Pract. 2014 Oct;68(10):1246-56. doi: 10.1111/ijcp.12443. Epub 2014 Apr 22. PMID 24754838
- [Derived] Chapple C, Sievert KD, MacDiarmid S, Khullar V, Radziszewski P, Nardo C, Thompson C, Zhou J, Haag-Molkenteller C. OnabotulinumtoxinA 100 U significantly improves all idiopathic overactive bladder symptoms and quality of life in patients with overactive bladder and urinary incontinence: a randomised, double-blind, placebo-controlled trial. Eur Urol. 2013 Aug;64(2):249-56. doi: 10.1016/j.eururo.2013.04.001. Epub 2013 Apr 10. PMID 23608668

RESULTS

PARTICIPANT FLOW:
Period: Treatment Cycle 1
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Started | 277 | 271
Completed | 257 | 247
Not Completed | 20 | 24
Period: Treatment Cycle 2
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Started | 163 (Not all participants who completed Treatment Cycle 1 went onto Treatment Cycle 2) | 223 (Not all participants who completed Treatment Cycle 1 went onto Treatment Cycle 2)
Completed | 156 | 215
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA | Total
Number analyzed (Participants) | 277 | 271 | 548
Age, Customized [Number; unit: Participants]
  < 40 years | 38 | 24 | 62
  Between 40 and 64 years | 115 | 139 | 254
  Between 65 and 74 years | 82 | 73 | 155
  ≥ 75 years | 42 | 35 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 229 | 473
  Male | 33 | 42 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Daily Episodes of Urinary Incontinence
Description: A urinary incontinence episode is defined as an incident of involuntary loss of urine as recorded in a patient bladder diary during the 3 days before the Baseline and Week 12 study visits. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: Incontinence episodes
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 277 | 271
Incontinence episodes
  Baseline | 5.52 (3.753) | 5.70 (3.858)
  Change from Baseline at Week 12 | -2.95 (3.576) | -1.03 (3.004)

2. Secondary Outcome: Change From Baseline in Number of Daily Micturition Episodes
Description: The number of micturition episodes (the number of times a patient urinates into the toilet) was recorded by the patient in a bladder diary during 3 consecutive days in the week prior to the Baseline and prior to the Week 12 study visit. A negative number change from baseline indicates a reduction in micturition episodes (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: micturition episodes
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 277 | 271
micturition episodes
  Baseline | 12.01 (4.007) | 11.77 (3.648)
  Change from Baseline at Week 12 | -2.56 (3.351) | -0.83 (2.523)

3. Secondary Outcome: Change From Baseline in Volume Voided Per Micturition
Description: The total volume voided was measured over one 24-hour period in the week prior to the Baseline and Week 12 study visit and recorded by the patient in the bladder diary. This was used to calculate volume voided per micturition. A positive number change from baseline indicates an increase in volume voided per micturition (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 277 | 271
milliliters
  Baseline | 144.2 (57.54) | 152.5 (59.27)
  Change from Baseline at Week 12 | 43.0 (65.27) | 12.6 (52.01)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were treated. S(AE)s are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 17/274 | 15/270
Other Adverse Events (participants affected / at risk) | 115/274 | 47/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA (N=274) | Placebo/onabotulinumtoxinA (N=270)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Vaginal disorder (Reproductive system and breast disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA (N=274) | Placebo/onabotulinumtoxinA (N=270)
Urinary tract infection (Infections and infestations) | 66 | 26
Bacteriuria (Infections and infestations) | 17 | 9
Dysuria (Renal and urinary disorders) | 16 | 11
Urinary retention (Renal and urinary disorders) | 16 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.